CLINICAL TRIAL: NCT05984381
Title: Efficacy and Safety of add-on Dapsone Versus add-on Methotrexate in Patients With Bullous Pemphigoid: A Randomized Controlled Trial
Brief Title: Efficacy and Safety of add-on Dapsone Versus add-on Methotrexate in Patients With Bullous Pemphigoid
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: All India Institute of Medical Sciences, Bhubaneswar (Other)
Responsible Party: Principal Investigator, Dr. Monalisa Jena, M.D., Additional Professor, All India Institute of Medical Sciences, Bhubaneswar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIIMS BBSR/PG Thesis/2023-24
Record Dates: First submitted 2023-07-24; First posted 2023-08-09 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Bullous Pemphigoid
Keywords: Bullous pemphigoid; Methotrexate; Dapsone; BP180; Blister; Erosions
MeSH Terms: conditions — Pemphigoid, Bullous; Blister | interventions — Prednisolone; Dapsone; Methotrexate

STUDY DESIGN:
Intervention Model Description: randomized, add-on, active-controlled, open-label, parallel-design clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prednisolone and Methotrexate (Control Arm) (Active Comparator): prednisolone 0.75mg/kg/day (a maximum dose of 40mg at baseline) and Methotrexate 15 mg weekly for 16 weeks.
  Interventions: Drug: Prednisolone; Drug: Methotrexate
- Prednisolone and Dapsone (Test Arm) (Experimental): prednisolone 0.75mg/kg/day (a maximum dose of 40mg at baseline) and Dapsone 100 mg/day for 16 weeks
  Interventions: Drug: Prednisolone; Drug: Dapsone

INTERVENTIONS:
Drug: Prednisolone — prednisolone 0.75mg/kg/day (a maximum dose of 40mg at baseline) orally
Drug: Dapsone — Dapsone 100 mg/day
  Arms: Prednisolone and Dapsone (Test Arm)
Drug: Methotrexate — Methotrexate 15 mg weekly
  Arms: Prednisolone and Methotrexate (Control Arm)

SUMMARY:
Bullous pemphigoid (BP) is an autoimmune subepidermal blistering disorder most commonly affecting the older population between 60-80 years old. The characteristic feature of BP is itchy patches associated with blisters and erosions. BP significantly affects the patient's quality of life as it causes physical discomfort with itchy patches, blisters, and erosions. Several pieces of evidence from previous studies showed that the production of autoantibodies against the hemidesmosomal anchoring proteins BP180 (Bullous Pemphigoid antigen (BPAG 2)) and BP230 (BPAG 1) is the most common cause for bullous pemphigoid.

Therapeutic latency, lack of efficacy in many patients, and adverse drug reactions are the primary concerns in the current bullous pemphigoid treatment paradigm, including high-dose steroid treatment. To overcome these treatment challenges, combination therapy with agents having a steroid-sparing effect like mycophenolate mofetil, cyclophosphamide, azathioprine, and Methotrexate are tested as an add-on to low-dose steroids. 8So other immunosuppressive agents with better safety profiles and more efficacy, like Dapsone and Methotrexate as an add-on to low-dose steroids, can be used.

Investigator's literature search found no randomized controlled trial with Dapsone versus Methotrexate as an add-on to first-line steroid has been conducted to compare the efficacy and safety in bullous pemphigoid patients. So, a randomized controlled trial has been planned to evaluate the safety and efficacy of add-on methotrexate versus Dapsone in bullous pemphigoid patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 of either sex with the clinical diagnosis of Bullous pemphigoid.
* Patients with BPDAI score ≥ 20 (moderate and severe BP).
* Patients must have characteristic clinical features of bullous pemphigoid at the screening and baseline visits. (Urticaria, bullae, pruritis).
* Patients who are willing to give informed written consent.

Exclusion Criteria:

* Patients on any steroid-sparing agents within one month of recruitment.
* Treatment with a systemic corticosteroid, sulfones, within the last week.
* Patients with Glucose 6 phosphate dehydrogenase deficiency.
* Decreased liver or renal function (creatinine > 2.0mg/dl, total bilirubin > 2.5 mg/dl).
* Severe acute infection, severe diabetes mellitus, untreated glaucoma, congenital or acquired immunodeficiency, active gastroduodenal ulcer, severe osteoporosis, severe cardiac disease (NYHA grade IV), MI in the last four weeks, severe schizophrenia or depression.
* Malignancies treated by cytotoxic or immunosuppressive medications.
* Anaemia (Hb <9 gm/dl), leucopenia (< 3 ×10 9 cells /L) or thrombocytopenia (< 100 × 10 9 cells/ L), and H/O porphyria.
* Patient with a history of hypersensitivity to Methotrexate or Dapsone.
* Vaccination in the last two weeks.
* Patients with HIV, Hepatitis B, and C infection.
* Pregnancy and lactation, women of childbearing age without effective contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-01-03 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
change in BPDAI (Bullous Pemphigoid Disease Area Index) score | 8 weeks and 16 weeks
  change in BPDAI (Bullous Pemphigoid Disease Area Index) score after treatment with prednisolone and methotraxate Vs Prednisolone and dapsone Score range from 0-360 (Minimum 0 and maximum 360) higher scores indicating greater disease activity

SECONDARY OUTCOMES:
change in serum BP180 | 16 weeks
  change in serum BP180 after treatment with prednisolone and methotraxate Vs Prednisolone and dapsone
the remission rate | 8 weeks and 16 weeks
  remission is defined as complete subsidence of all lesions without prednisolone or minimal prednisolone dose of 10 mg or less
the cumulative prednisolone dose | 16 weeks
  cumulative prednisolone dose after treatment with prednisolone and methotraxate Vs Prednisolone and dapsone
time to the initial flare | 16 weeks
  time to the initial flare after treatment with prednisolone and methotraxate Vs Prednisolone and dapsone
number of flares in study groups | 16 weeks
  number of flares in study groups after treatment with prednisolone and methotraxate Vs Prednisolone and dapsone
change in the Dermatological life quality index (DLQI) | 8 weeks and 16 weeks
  change in the Dermatological life quality index (DLQI) after treatment with prednisolone and methotraxate Vs Prednisolone and dapsone maximum of 30 and a minimum of 0 The higher the score, the more quality of life is impaired.
treatment-emergent adverse events | 16 weeks
  treatment-emergent adverse events in both the groups

CONTACTS AND LOCATIONS:
Overall Officials: Rituparna Maiti, MD, Study Director — Professor
Locations (1):
- AIIMS Bhubaneswar, Bhubaneswar, Odisha, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lu L, Chen L, Xu Y, Liu A. Global incidence and prevalence of bullous pemphigoid: A systematic review and meta-analysis. J Cosmet Dermatol. 2022 Oct;21(10):4818-4835. doi: 10.1111/jocd.14797. Epub 2022 Feb 1. PMID 35080093
- [Background] Chen X, Zhang Y, Luo Z, Wu Y, Niu T, Zheng J, Xie Y. Prognostic factors for mortality in bullous pemphigoid: A systematic review and meta-analysis. PLoS One. 2022 Apr 15;17(4):e0264705. doi: 10.1371/journal.pone.0264705. eCollection 2022. PMID 35427358
- [Background] Genovese G, Di Zenzo G, Cozzani E, Berti E, Cugno M, Marzano AV. New Insights Into the Pathogenesis of Bullous Pemphigoid: 2019 Update. Front Immunol. 2019 Jul 2;10:1506. doi: 10.3389/fimmu.2019.01506. eCollection 2019. PMID 31312206
- [Background] Patton T, Korman N. Role of methotrexate in the treatment of bullous pemphigoid in the elderly. Drugs Aging. 2008;25(8):623-9. doi: 10.2165/00002512-200825080-00001. PMID 18665656
- [Background] Tirado-Sanchez A, Diaz-Molina V, Ponce-Olivera RM. Efficacy and safety of azathioprine and dapsone as an adjuvant in the treatment of bullous pemphigoid. Allergol Immunopathol (Madr). 2012 May-Jun;40(3):152-5. doi: 10.1016/j.aller.2010.12.009. Epub 2011 Apr 14. PMID 21497011
- [Background] Sticherling M, Franke A, Aberer E, Glaser R, Hertl M, Pfeiffer C, Rzany B, Schneider S, Shimanovich I, Werfel T, Wilczek A, Zillikens D, Schmidt E. An open, multicentre, randomized clinical study in patients with bullous pemphigoid comparing methylprednisolone and azathioprine with methylprednisolone and dapsone. Br J Dermatol. 2017 Nov;177(5):1299-1305. doi: 10.1111/bjd.15649. Epub 2017 Oct 29. PMID 28494097
- [Background] Rashid H, Lamberts A, Diercks GFH, Pas HH, Meijer JM, Bolling MC, Horvath B. Oral Lesions in Autoimmune Bullous Diseases: An Overview of Clinical Characteristics and Diagnostic Algorithm. Am J Clin Dermatol. 2019 Dec;20(6):847-861. doi: 10.1007/s40257-019-00461-7. PMID 31313078
- [Background] Reunala T, Salmi TT, Hervonen K. Dermatitis herpetiformis: pathognomonic transglutaminase IgA deposits in the skin and excellent prognosis on a gluten-free diet. Acta Derm Venereol. 2015 Nov;95(8):917-22. doi: 10.2340/00015555-2162. PMID 26059085